CLINICAL TRIAL: NCT01302080
Title: SPRITES: SERTRALINE PEDIATRIC REGISTRY FOR THE EVALUATION OF SAFETY A NON-INTERVENTIONAL, LONGITUDINAL, COHORT STUDY TO EVALUATE THE EFFECTS OF LONG-TERM SERTRALINE TREATMENT IN CHILDREN AND ADOLESCENTS
Brief Title: Sertraline Pediatric Registry for the Evaluation of Safety (SPRITES)
Acronym: SPRITES
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0501093; SPRITES (Other: Alias Study Number)
Record Dates: First submitted 2011-02-01; First posted 2011-02-23 (Estimated); Results first posted 2021-10-08 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Obsessive Compulsive Disorder
Keywords: prospective; cohort; sertraline; long-term impact; cognition; emotional and physical development; pubertal maturation
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Sertraline; Psychotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sertraline-treated: enrolled subjects beginning treatment for one of the study qualifying disorders with sertraline
  Interventions: Drug: sertraline
- psychotherapy only: enrolled subjects beginning treatment for one of the study qualifying disorders with psychotherapy
  Interventions: Behavioral: psychotherapy

INTERVENTIONS:
Drug: sertraline — Non interventional study - drug, dose, duration etc as per USPI and clinician discretion
  Groups: Sertraline-treated
Behavioral: psychotherapy — Non-interventional study- as above
  Groups: psychotherapy only

SUMMARY:
To evaluate the long-term impact of treatment with sertraline on aspects of cognitive, emotional and physical development and pubertal maturation in pediatric subjects ages 6 to 16 years (inclusive) with a diagnosis of anxiety disorder, depressive disorder or obsessive compulsive disorder.

DETAILED DESCRIPTION:
Purposive sample: patients are not randomly selected, that is, he or she must meet certain inclusion criteria in order to qualify as a potential study participant.

ELIGIBILITY:
Inclusion Criteria:

* Children age 6 to 16 (inclusive) with anxiety, depression, or obsessive-compulsive disorder, receiving treatment in outpatient setting, and who are prescribed a new prescription for sertraline to treat one of the above study-qualifying disorders or beginning psychotherapy for same.

Exclusion Criteria:

* Psychotic at study entry
* Diagnosis of bipolar disorder
* Diagnosis of schizoaffective or schizophrenia
* Anorexia
* Bulimia or eating disorder not otherwise specified (NOS)
* Autism
* Pervasive developmental disorder
* High risk of suicide within 2 weeks of initiating study treatment
* Significant mental retardation
* Taking an antidepressant medication other than sertraline, first or second generation antipsychotic, lithium, psychostimulant

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The accessible population is children meeting inclusion/exclusion criteria from US centers in various clinical settings, including the Child and Adolescent Psychiatry Trials Network (CAPTN). From these, the study-eligible population (all children age 6 to 16 (inclusive) with an anxiety, depressive, or obsessive-compulsive disorder, who are exposed to sertraline under real-world conditions) will comprise an inception cohort of enrolled subjects beginning treatment for one of the study-qualifying disorders with sertraline or psychotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 941 (Actual)
Dates: Start 2012-04-04 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (44):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Sun Valley Research Center, Imperial, California
  - UCLA Semel institute, Los Angeles, California
  - Institute of Living/Hartford Hospital, Hartford, Connecticut
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - University of Florida, Gainesville, Florida
  - Nemours Children's Clinic, Dept. of Psychology and Psychiatry, Jacksonville, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Harmonex Neuroscience of Pensacola, Pensacola, Florida
  - University of South Florida - Rothman Center, St. Petersburg, Florida
  - Georgia Regents University Augusta, Augusta, Georgia
  - Institute for Behavioral Medicine, LLC, Smyrna, Georgia
  - Family Behavioral Health, Plainfield, Illinois
  - University of Kansas School of Medicine/Dept. of Psychiatry, Kansas City, Kansas
  - Family Service and Guidance Center, Topeka, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Neuroscientific Insights, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Debora A. LaMonica, MD, South Yarmouth, Massachusetts
  - Baystate Medical Center, Child Behavioral Health Research, Springfield, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Comprehensive Psychiatric Associates, Gladstone, Missouri
  - Saint John's Clinic, Springfield, Missouri
  - Jersey Shore University Medical Center/Meridian Health, Neptune City, New Jersey
  - Children's Specialized Hospital, Toms River, New Jersey
  - Finger Lakes Clinical Research, Rochester, New York
  - 3-C Family Services, P.A., Cary, North Carolina
  - Duke University Medical Center, Division of Child & Adolescent Psychiatry, Durham, North Carolina
  - Scott George Crowder, M.D., Wilmington, North Carolina
  - Family Center by the Falls, Chagrin Falls, Ohio
  - University Of Cincinnati, Cincinnati, Ohio
  - Cincinnati Childrens Hospital and Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Department of Psychiatry Child/Adolescent, Cleveland, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Child Guidance Resource Center, Havertown, Pennsylvania
  - Tullahoma Pediatrics PLLC, Tullahoma, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Bay Pointe Behavioral Health Service, Inc., Friendswood, Texas
  - Midtown Psychiatry and TMS Center, Houston, Texas
  - Peter Ly MD, Houston, Texas
  - Focus and Balance, LLC, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Clinical Research Partners, LLC, Petersburg, Virginia
  - McLean Hospital - Harvard Medical School, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Kolitsopoulos F, Ramaker S, Compton SN, Broderick S, Orazem J, Bao W, Lokhnygina Y, Marschall K, Chappell P. Effects of Long-Term Sertraline Use on Pediatric Growth and Development: The Sertraline Pediatric Registry for The Evaluation of Safety (SPRITES). J Child Adolesc Psychopharmacol. 2023 Feb;33(1):2-13. doi: 10.1089/cap.2022.0048. PMID 36799958
- [Derived] Kolitsopoulos F, Ramaker S, Compton S, Broderick S, Orazem J, Bao W, Lokhnygina Y, Chappell P. Sertraline Pediatric Registry for the Evaluation of Safety: Design and Clinical Characteristics of Pediatric Patients Prescribed Sertraline. J Child Adolesc Psychopharmacol. 2021 Aug;31(6):411-420. doi: 10.1089/cap.2020.0170. Epub 2021 Jul 21. PMID 34287023
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0501093&StudyName=Sertraline%20Pediatric%20Registry%20for%20the%20Evaluation%20of%20Safety%20%28SPRITES%29%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional observational study. Participants to be enrolled were of age 6 to 16 (inclusive), exposed to sertraline (with or without psychotherapy) and exposed to psychotherapy alone under real world conditions. Participants exposed and unexposed to sertraline were followed for a maximum of 3 years.
Pre-assignment Details: Participants switched from 1 treatment to another throughout the study, irrespective in which arm they were enrolled. Hence, number of participants for reporting arms were different at different visits.
Groups:
- Sertraline: Participants at Baseline (Day 1) or within 45 days of enrollment, initiated treatment with sertraline in routine clinical settings according to United States prescribing information (USPI) provided by their physician. Participants in this group were on sertraline only or sertraline and any other treatment. Treatment here was the one which was planned for the participants at baseline.
- Psychotherapy: Participants, 1) who were not taking sertraline or who failed a trial of sertraline judged adequate in dose and duration, and 2) initiated psychosocial/psychotherapy rather than pharmacological treatment on or within 45 days of enrollment, for the same spectrum of mental health conditions that could have been treated with a selective serotonin reuptake inhibitor (SSRI) medication. Participants in this group were on psychotherapy only or no treatment at all.
Period: Overall Study
Arm/Group | Sertraline | Psychotherapy
Started | 696 (Out of 696 participants, 1 participant started treatment with another antidepressant alone or along with psychotherapy.) | 245 (Out of 245 participants, 2 participants started treatment with another antidepressant alone or along with psychotherapy.)
Completed | 330 | 102
Not Completed | 366 | 143
Not completed — Withdrew Consent | 92 | 39
Not completed — Patient/Family Moved | 28 | 3
Not completed — Lost to Follow-up | 192 | 93
Not completed — Death | 1 | 0
Not completed — Other | 52 | 8
Not completed — Reason Missing For Discontinuation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants in the database who had informed consent.
Groups:
- Sertraline: Participants at Baseline (Day 1) or within 45 days of enrollment, initiated treatment with sertraline in routine clinical settings according to USPI provided by their physician.
- Other Antidepressant: Use of other antidepressants at baseline was a study exclusion criterion, however, a few participants were enrolled who initiated treatment with an antidepressant.
- Psychotherapy: Participants, 1) who were not taking sertraline or who failed a trial of sertraline judged adequate in dose and duration, and 2) initiated psychosocial rather than pharmacological treatment on or within 45 days of enrollment, for the same spectrum of mental health conditions that could have been treated with a SSRI medication.
- Total: Total of all reporting groups
Arm/Group | Sertraline | Other Antidepressant | Psychotherapy | Total
Number analyzed (Participants) | 695 | 3 | 243 | 941
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (2.9) | 14.0 (3.0) | 11.0 (2.9) | 11.9 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 405 | 3 | 130 | 538
  Male | 290 | 0 | 113 | 403
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 73 | 1 | 24 | 98
  Not Hispanic or Latino | 622 | 2 | 219 | 843
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 23 | 0 | 2 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 66 | 0 | 15 | 81
  White | 588 | 3 | 208 | 799
  More than one race | 14 | 0 | 13 | 27
  Unknown or Not Reported | 4 | 0 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cognitive Function Using Trails B at Month 3
Description: Trail B test is a set of shifting task, in which participants were asked to drawn a line from number 1 to letter A, then to number 2, then to letter B, then to number 3, then to letter C then so forth until they connected the circles as quickly as possible, without lifting pen or pencil from the paper. Participant was timed (maximum time limit was 300 seconds or 5 minutes) to connect the "trail." If the participant made an error, and it was pointed out immediately, the participant was allowed to correct it. Errors affected the participant's score only in that the correction of errors was included in the completion time for the task. A higher number of errors was indicative of a higher cognitive deficit. Raw results were the number of seconds required to complete the task; therefore, higher scores reveal greater impairment. Raw results based on age norms were transformed to Z-scores. Z-score = actual value minus normative value divided by standard deviation.
Time Frame: Baseline, Month 3
Population: Analysis population included all participants in the database who had informed consent. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Sertraline: At baseline, participants in this group were those at Baseline (Day 1) or within 45 days of enrollment, initiated treatment with sertraline in routine clinical settings according to USPI provided by their physician.
  At a visit post baseline, participants in this group were on sertraline only or sertraline and any other treatment since the previous visit.
- Other Antidepressants: At baseline, use of other antidepressants at baseline was a study exclusion criterion. However, a few participants were enrolled and initiated treatment with an antidepressant other than sertraline, and hence included in this group. At a visit post baseline, participants in this group were on another antidepressant only or on another antidepressant and psychotherapy since the previous visit.
- Psychotherapy: At baseline, participants in this group were on psychotherapy only and were those who 1) were not taking sertraline or who failed a trial of sertraline judged adequate in dose and duration, and 2) initiated psychosocial rather than pharmacological treatment on or within 45 days of enrollment, for the same spectrum of mental health conditions that could have been treated with a SSRI medication. At a visit post baseline, participants in this group were those on psychotherapy only or no treatment at all since the previous visit.
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 666 | 3 | 224
Z-score
  Baseline | 1.03 (2.3) | 1.23 (1.0) | 0.61 (1.8)
  Change at Week 3: number analyzed (Participants) | 527 | 3 | 163
  Change at Week 3 | -0.39 (1.6) | -0.09 (0.5) | -0.03 (2.3)

2. Primary Outcome: Change From Baseline in Cognitive Function Using Trails B at Month 6
Description: as for outcome 1
Time Frame: Baseline, Month 6
Population: Analysis population included all participants in the database who had informed consent. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 460 | 35 | 159
Z-score | -0.64 (2.2) | -0.65 (1.0) | -0.16 (1.9)

3. Primary Outcome: Change From Baseline in Cognitive Function Using Trails B at Month 12
Description: as for outcome 1
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 367 | 57 | 138
Z-score | -0.72 (2.3) | -0.22 (1.4) | -0.27 (2.4)

4. Primary Outcome: Change From Baseline in Cognitive Function Using Trails B at Month 18
Description: as for outcome 1
Time Frame: Baseline, Month 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 290 | 70 | 138
Z-score | -0.57 (1.9) | -0.65 (2.2) | -0.22 (2.8)

5. Primary Outcome: Change From Baseline in Cognitive Function Using Trails B at Month 24
Description: as for outcome 1
Time Frame: Baseline, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 247 | 70 | 134
Z-score | -0.44 (2.2) | -1.08 (1.7) | -0.18 (3.4)

6. Primary Outcome: Change From Baseline in Cognitive Function Using Trails B at Month 30
Description: as for outcome 1
Time Frame: Baseline, Month 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 209 | 63 | 141
Z-score | -0.74 (2.1) | -0.61 (2.4) | -0.18 (4.2)

7. Primary Outcome: Change From Baseline in Cognitive Function Using Trails B at Month 36
Description: as for outcome 1
Time Frame: Baseline, Month 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 193 | 56 | 154
Z-score | -0.25 (2.9) | -0.13 (3.6) | -0.59 (2.6)

8. Primary Outcome: Change From Baseline in Cognitive Function Using Metacognition Index From Behavior Rating Inventory of Executive Function (BRIEF) at Month 3
Description: BRIEF has 86-items to measure the neurocognitive performance for 8 subscales: inhibit, shift, emotional control, initiate, working memory, plan-organize, organization of materials and monitor. These are subsumed in 2 broad factors: a behavior regulation index consisted inhibit, shift, and emotional control subscales, a metacognition index consisted working memory, initiate, plan/organize, organization of materials, and task-monitor scale. Each item had a 3-point scale (1= never, 2= sometimes, 3= often). Z-score was based on mean raw score for T-score= 50 and SD = +/- 10. (actual value raw score at T=50)/SD (mean SD where T=40,60), based on age and gender norms from BRIEF professional manual. T-score provided information of individual's scores relative to scores of respondents in the standardization sample. Lower Z- scores indicated better functioning.
Time Frame: Baseline, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 686 | 3 | 237
Z-score
  Baseline | 62.93 (11.3) | 57.67 (5.5) | 59.27 (13.0)
  Change at Week 3: number analyzed (Participants) | 539 | 2 | 170
  Change at Week 3 | -2.29 (7.8) | 4.50 (13.4) | -1.88 (7.3)

9. Primary Outcome: Change From Baseline in Cognitive Function Using Metacognition Index From Behavior Rating Inventory of Executive Function (BRIEF) at Month 6
Description: as for outcome 8
Time Frame: Baseline, Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 467 | 35 | 166
Z-score | -2.53 (8.8) | -1.54 (8.8) | -2.74 (8.7)

10. Primary Outcome: Change From Baseline in Cognitive Function Using Metacognition Index From Behavior Rating Inventory of Executive Function (BRIEF) at Month 12
Description: as for outcome 8
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 370 | 58 | 140
Z-score | -3.12 (9.1) | -1.97 (8.3) | -2.81 (9.0)

11. Primary Outcome: Change From Baseline in Cognitive Function Using Metacognition Index From Behavior Rating Inventory of Executive Function (BRIEF) at Month 18
Description: as for outcome 8
Time Frame: Baseline, Month 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 290 | 69 | 140
Z-score | -2.40 (9.2) | -1.57 (9.9) | -3.13 (8.3)

12. Primary Outcome: Change From Baseline in Cognitive Function Using Metacognition Index From Behavior Rating Inventory of Executive Function (BRIEF) at Month 24
Description: as for outcome 8
Time Frame: Baseline, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 248 | 66 | 133
Z-score | -3.37 (10.0) | -3.14 (9.0) | -4.16 (9.5)

13. Primary Outcome: Change From Baseline in Cognitive Function Using Metacognition Index From Behavior Rating Inventory of Executive Function (BRIEF) at Month 30
Description: as for outcome 8
Time Frame: Baseline, Month 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 200 | 59 | 135
Z-score | -3.60 (11.2) | -4.39 (8.7) | -4.53 (10.2)

14. Primary Outcome: Change From Baseline in Cognitive Function Using Metacognition Index From Behavior Rating Inventory of Executive Function (BRIEF) at Month 36
Description: as for outcome 8
Time Frame: Baseline, Month 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 184 | 54 | 141
Z-score | -3.96 (12.1) | -3.87 (10.4) | -4.62 (10.9)

15. Primary Outcome: Change From Baseline in Behavioral/Emotional Regulation Using the Behavior Regulation Index From BRIEF at Month 3
Description: as for outcome 8
Time Frame: Baseline, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 692 | 3 | 238
Z-score
  Baseline | 65.15 (12.0) | 58.67 (4.0) | 61.88 (12.6)
  Change at Week 3: number analyzed (Participants) | 544 | 2 | 171
  Change at Week 3 | -3.08 (9.1) | -1.50 (0.7) | -2.39 (7.4)

16. Primary Outcome: Change From Baseline in Behavioral/Emotional Regulation Using the Behavior Regulation Index From BRIEF at Month 6
Description: as for outcome 8
Time Frame: Baseline, Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 472 | 36 | 167
Z-score | -4.06 (9.4) | -3.14 (9.7) | -3.62 (8.9)

17. Primary Outcome: Change From Baseline in Behavioral/Emotional Regulation Using the Behavior Regulation Index From BRIEF at Month 12
Description: as for outcome 8
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 373 | 59 | 140
Z-score | -5.42 (10.1) | -2.44 (8.2) | -5.01 (9.5)

18. Primary Outcome: Change From Baseline in Behavioral/Emotional Regulation Using the Behavior Regulation Index From BRIEF at Month 18
Description: as for outcome 8
Time Frame: Baseline, Month 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 294 | 71 | 140
Z-score | -5.21 (9.9) | -3.59 (9.9) | -4.48 (9.2)

19. Primary Outcome: Change From Baseline in Behavioral/Emotional Regulation Using the Behavior Regulation Index From BRIEF at Month 24
Description: as for outcome 8
Time Frame: Baseline, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 252 | 68 | 133
Z-score | -6.21 (11.2) | -5.78 (8.8) | -6.05 (9.9)

20. Primary Outcome: Change From Baseline in Behavioral/Emotional Regulation Using the Behavior Regulation Index From BRIEF at Month 30
Description: as for outcome 8
Time Frame: Baseline, Month 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 204 | 61 | 136
Z-score | -6.92 (10.8) | -5.23 (10.0) | -6.53 (10.4)

21. Primary Outcome: Change From Baseline in Behavioral/Emotional Regulation Using the Behavior Regulation Index From BRIEF at Month 36
Description: as for outcome 8
Time Frame: Baseline, Month 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 188 | 55 | 142
Z-score | -7.44 (11.1) | -7.24 (10.6) | -6.22 (11.2)

22. Primary Outcome: Change From Baseline in Height at Month 3
Description: Height was measured and referenced to norms according to standardized procedures from the national health and nutrition examination survey (NHANES III). Raw height measurements were norm-adjusted transformed to Z-score using formula: Z-score= actual value minus normative value divided by standard deviation based on centers for disease control (CDC) norms for age and gender.
Time Frame: Baseline, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 693 | 3 | 243
Z-score
  Baseline | 0.31 (1.1) | 0.76 (1.4) | 0.32 (1.1)
  Change at Month 3: number analyzed (Participants) | 554 | 3 | 174
  Change at Month 3 | 0.00 (0.3) | -0.03 (0.1) | -0.01 (0.3)

23. Primary Outcome: Change From Baseline in Height at Month 6
Description: Height was measured and referenced to norms according to standardized procedures from the national health and nutrition examination survey (NHANES III). Raw height measurements were norm-adjusted transformed to Z-score using formula: Z-score= actual value minus normative value divided by standard deviation based on CDC norms for age and gender.
Time Frame: Baseline, Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 478 | 36 | 170
Z-score | -0.02 (0.3) | 0.07 (0.4) | 0.00 (0.4)

24. Primary Outcome: Change From Baseline in Height at Month 12
Description: as for outcome 23
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 381 | 59 | 144
Z-score | -0.01 (0.4) | 0.06 (0.5) | -0.04 (0.4)

25. Primary Outcome: Change From Baseline in Height at Month 18
Description: as for outcome 23
Time Frame: Baseline, Month 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 305 | 74 | 145
Z-score | -0.03 (0.5) | 0.00 (0.5) | -0.02 (0.6)

26. Primary Outcome: Change From Baseline in Height at Month 24
Description: as for outcome 23
Time Frame: Baseline, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 263 | 70 | 138
Z-score | 0.01 (0.5) | -0.02 (0.6) | -0.02 (0.5)

27. Primary Outcome: Change From Baseline in Height at Month 30
Description: as for outcome 23
Time Frame: Baseline, Month 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 218 | 66 | 148
Z-score | 0.01 (0.7) | -0.10 (0.6) | 0.00 (0.6)

28. Primary Outcome: Change From Baseline in Height at Month 36
Description: as for outcome 23
Time Frame: Baseline, Month 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 203 | 62 | 160
Z-score | 0.00 (0.7) | -0.04 (0.7) | -0.02 (0.9)

29. Primary Outcome: Change From Baseline in Weight at Month 3
Description: Weight was measured and referenced to norms according to standardized procedures from the national health and nutrition examination survey (NHANES III). Raw weight measurements were norm-adjusted transformed to Z-score using formula: Z-score= actual value minus normative value divided by standard deviation based on CDC norms for age and gender.
Time Frame: Baseline, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 693 | 3 | 243
Z-score
  Baseline | 0.58 (1.2) | 0.88 (0.7) | 0.42 (1.0)
  Change at Month 3: number analyzed (Participants) | 554 | 3 | 173
  Change at Month 3 | 0.02 (0.2) | -0.22 (0.1) | -0.03 (0.2)

30. Primary Outcome: Change From Baseline in Weight at Month 6
Description: as for outcome 29
Time Frame: Baseline, Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 478 | 36 | 170
Z-score | 0.03 (0.3) | 0.01 (0.3) | -0.05 (0.3)

31. Primary Outcome: Change From Baseline in Weight at Month 12
Description: as for outcome 29
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 382 | 59 | 144
Z-score | 0.10 (0.4) | 0.06 (0.5) | 0.00 (0.4)

32. Primary Outcome: Change From Baseline in Weight at Month 18
Description: as for outcome 29
Time Frame: Baseline, Month 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 305 | 74 | 145
Z-score | 0.14 (0.5) | 0.07 (0.6) | -0.01 (0.5)

33. Primary Outcome: Change From Baseline in Weight at Month 24
Description: as for outcome 29
Time Frame: Baseline, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 263 | 70 | 138
Z-score | 0.16 (0.5) | 0.15 (0.6) | 0.00 (0.6)

34. Primary Outcome: Change From Baseline in Weight at Month 30
Description: as for outcome 29
Time Frame: Baseline, Month 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 218 | 66 | 148
Z-score | 0.16 (0.6) | 0.11 (0.6) | 0.04 (0.6)

35. Primary Outcome: Change From Baseline in Weight at Month 36
Description: as for outcome 29
Time Frame: Baseline, Month 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 203 | 62 | 162
Z-score | 0.17 (0.6) | 0.17 (0.7) | 0.02 (0.6)

36. Primary Outcome: Change From Baseline in Body Mass Index (BMI) at Month 3
Description: BMI is participant's weight in kilograms divided by the square of height in meters. BMI was measured and referenced to norms according to standardized procedures from the national health and nutrition examination survey (NHANES III). Raw BMI measurements were norm-adjusted transformed to Z-score using formula: Z-score = actual value minus normative value divided by standard deviation based on CDC norms for age and gender.
Time Frame: Baseline, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 693 | 3 | 243
Z-score
  Baseline | 0.48 (1.3) | 0.79 (0.4) | 0.27 (1.3)
  Change at Month 3: number analyzed (Participants) | 554 | 3 | 173
  Change at Month 3 | 0.02 (0.3) | -0.26 (0.2) | -0.03 (0.3)

37. Primary Outcome: Change From Baseline in Body Mass Index (BMI) at Month 6
Description: as for outcome 36
Time Frame: Baseline, Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 478 | 36 | 170
Z-score | 0.04 (0.4) | -0.03 (0.4) | -0.06 (0.4)

38. Primary Outcome: Change From Baseline in Body Mass Index (BMI) at Month 12
Description: as for outcome 36
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 381 | 59 | 144
Z-score | 0.13 (0.5) | 0.06 (0.6) | 0.04 (0.6)

39. Primary Outcome: Change From Baseline in Body Mass Index (BMI) at Month 18
Description: as for outcome 36
Time Frame: Baseline, Month 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 305 | 74 | 145
Z-score | 0.18 (0.6) | 0.07 (0.8) | -0.04 (0.6)

40. Primary Outcome: Change From Baseline in Body Mass Index (BMI) at Month 24
Description: as for outcome 36
Time Frame: Baseline, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 263 | 70 | 138
Z-score | 0.17 (0.7) | 0.20 (0.9) | -0.01 (0.7)

41. Primary Outcome: Change From Baseline in Body Mass Index (BMI) at Month 30
Description: as for outcome 36
Time Frame: Baseline, Month 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 218 | 66 | 148
Z-score | 0.16 (0.8) | 0.15 (0.8) | 0.03 (0.7)

42. Primary Outcome: Change From Baseline in Body Mass Index (BMI) at Month 36
Description: as for outcome 36
Time Frame: Baseline, Month 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 203 | 62 | 160
Z-score | 0.17 (0.8) | 0.21 (0.9) | 0.01 (0.7)

43. Primary Outcome: Primary: Number of Participants With Tanner Staging Evaluation at Baseline: All Males
Description: Tanner stage defines physical measurements of development based on external primary and secondary sex characteristics. The physical changes for males in pubertal development (pubic hair, penis and testes) were assessed. Participants were evaluated for genital development, with values ranging from stage 1 (pre-pubertal characteristics) to stage 5 (adult or mature characteristics).
Time Frame: Baseline (prior to or within 45 Days of initiating treatment, if exposed) and after parental/guardian provided permission and assent
Population: Analysis population included all participants in the database who had informed consent. Here, "Overall Number of Participants Analyzed" signifies number of male participants evaluable for this outcome measure. There were no male participants in reporting arm "Other Antidepressant" at Baseline, hence no data collected and evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 288 | 0 | 113
Participants
  Stage 1 | 122 |  | 58
  Stage 2 | 53 |  | 20
  Stage 3 | 45 |  | 17
  Stage 4 | 53 |  | 15
  Stage 5 | 15 |  | 3

44. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 3: All Males
Description: as for outcome 43
Time Frame: Month 3
Population: Analysis population included all participants in the database who had informed consent. Here, "Overall Number of Participants Analyzed" signifies number of male participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 230 | 1 | 80
Participants
  Stage 1 | 94 | 1 | 42
  Stage 2 | 40 | 0 | 10
  Stage 3 | 43 | 0 | 14
  Stage 4 | 45 | 0 | 11
  Stage 5 | 8 | 0 | 3

45. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 6: All Males
Description: as for outcome 43
Time Frame: Month 6
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 203 | 14 | 77
Participants
  Stage 1 | 75 | 6 | 36
  Stage 2 | 44 | 2 | 11
  Stage 3 | 34 | 3 | 14
  Stage 4 | 43 | 2 | 14
  Stage 5 | 7 | 1 | 2

46. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 12: All Males
Description: as for outcome 43
Time Frame: Month 12
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 164 | 24 | 69
Participants
  Stage 1 | 55 | 7 | 30
  Stage 2 | 37 | 2 | 11
  Stage 3 | 26 | 5 | 12
  Stage 4 | 36 | 8 | 12
  Stage 5 | 10 | 2 | 4

47. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 18: All Males
Description: as for outcome 43
Time Frame: Month 18
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 136 | 33 | 57
Participants
  Stage 1 | 39 | 9 | 20
  Stage 2 | 31 | 5 | 11
  Stage 3 | 19 | 6 | 12
  Stage 4 | 33 | 7 | 9
  Stage 5 | 14 | 6 | 5

48. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 24: All Males
Description: as for outcome 43
Time Frame: Month 24
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 112 | 34 | 62
Participants
  Stage 1 | 32 | 7 | 13
  Stage 2 | 27 | 9 | 12
  Stage 3 | 17 | 6 | 14
  Stage 4 | 22 | 6 | 16
  Stage 5 | 14 | 6 | 7

49. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 30: All Males
Description: as for outcome 43
Time Frame: Month 30
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 86 | 33 | 64
Participants
  Stage 1 | 23 | 5 | 10
  Stage 2 | 18 | 7 | 8
  Stage 3 | 16 | 5 | 19
  Stage 4 | 15 | 6 | 19
  Stage 5 | 14 | 10 | 8

50. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 36: All Males
Description: as for outcome 43
Time Frame: Month 36
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 84 | 34 | 75
Participants
  Stage 1 | 18 | 6 | 7
  Stage 2 | 18 | 4 | 12
  Stage 3 | 14 | 10 | 15
  Stage 4 | 22 | 4 | 25
  Stage 5 | 12 | 10 | 16

51. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Baseline: All Females
Description: Tanner stage defines physical measurements of development based on external primary and secondary sex characteristics. The physical changes for females in pubertal development were assessed. Participants were evaluated for pubic hair distribution, breast development, with values ranging from stage 1 (pre-pubertal characteristics) to stage 5 (adult or mature characteristics).
Time Frame: as for outcome 43
Population: Analysis population included all participants in the database who had informed consent. Here, "Overall Number of Participants Analyzed" signifies number of female participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 401 | 3 | 130
Participants
  Stage 1 | 81 | 1 | 39
  Stage 2 | 40 | 0 | 21
  Stage 3 | 61 | 0 | 25
  Stage 4 | 146 | 1 | 28
  Stage 5 | 73 | 1 | 17

52. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 3: All Females
Description: as for outcome 51
Time Frame: Month 3
Population: as for outcome 51
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 323 | 2 | 94
Participants
  Stage 1 | 59 | 1 | 30
  Stage 2 | 37 | 0 | 13
  Stage 3 | 47 | 0 | 14
  Stage 4 | 108 | 0 | 24
  Stage 5 | 72 | 1 | 13

53. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 6: All Females
Description: as for outcome 51
Time Frame: Month 6
Population: as for outcome 51
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 275 | 22 | 91
Participants
  Stage 1 | 43 | 1 | 22
  Stage 2 | 31 | 4 | 13
  Stage 3 | 46 | 2 | 18
  Stage 4 | 90 | 10 | 18
  Stage 5 | 65 | 5 | 20

54. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 12: All Females
Description: as for outcome 51
Time Frame: Month 12
Population: as for outcome 51
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 218 | 35 | 75
Participants
  Stage 1 | 27 | 5 | 9
  Stage 2 | 27 | 2 | 15
  Stage 3 | 31 | 5 | 12
  Stage 4 | 71 | 11 | 24
  Stage 5 | 62 | 12 | 15

55. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 18: All Females
Description: as for outcome 51
Time Frame: Month 18
Population: as for outcome 51
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 169 | 40 | 88
Participants
  Stage 1 | 17 | 4 | 9
  Stage 2 | 14 | 2 | 14
  Stage 3 | 22 | 2 | 13
  Stage 4 | 57 | 14 | 31
  Stage 5 | 59 | 18 | 21

56. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 24: All Females
Description: as for outcome 51
Time Frame: Month 24
Population: as for outcome 51
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 151 | 37 | 76
Participants
  Stage 1 | 13 | 2 | 8
  Stage 2 | 15 | 3 | 10
  Stage 3 | 16 | 1 | 13
  Stage 4 | 49 | 11 | 24
  Stage 5 | 58 | 20 | 21

57. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 30: All Females
Description: as for outcome 51
Time Frame: Month 30
Population: as for outcome 51
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 132 | 33 | 84
Participants
  Stage 1 | 10 | 1 | 3
  Stage 2 | 15 | 2 | 9
  Stage 3 | 15 | 1 | 8
  Stage 4 | 34 | 8 | 29
  Stage 5 | 58 | 21 | 35

58. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 36: All Females
Description: as for outcome 51
Time Frame: Month 36
Population: as for outcome 51
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 120 | 30 | 88
Participants
  Stage 1 | 9 | 0 | 2
  Stage 2 | 9 | 2 | 9
  Stage 3 | 9 | 7 | 8
  Stage 4 | 32 | 7 | 25
  Stage 5 | 61 | 14 | 44

59. Secondary Outcome: Number of Participants in Each Category of Clinical Global Impression-Improvement (CGI-I) Scale at Month 3, 6, 12, 18, 24, 30 and 36
Description: CGI-I scale was a 7-point scale used to rate improvement in the participant's condition (benefits). Scale range/categories: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = Not changed, 5 = minimally worse, 6 = much worse, and 7 = very much worse. Higher score indicated worse condition.
Time Frame: Month 3, 6, 12, 18, 24, 30 and 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 556 | 73 | 176
Participants
  Month 3: number analyzed (Participants) | 556 | 3 | 176
  Month 3: Very Much Improved | 77 | 0 | 17
  Month 3: Much Improved | 223 | 0 | 51
  Month 3: Minimally Improved | 151 | 1 | 69
  Month 3: Not Changed | 63 | 1 | 29
  Month 3: Minimally Worse | 20 | 0 | 3
  Month 3: Much Worse | 21 | 0 | 5
  Month 3: Very Much Worse | 1 | 1 | 2
  Month 6: number analyzed (Participants) | 478 | 34 | 167
  Month 6: Very Much Improved | 96 | 2 | 29
  Month 6: Much Improved | 220 | 14 | 64
  Month 6: Minimally Improved | 87 | 7 | 48
  Month 6: Not Changed | 44 | 8 | 21
  Month 6: Minimally Worse | 15 | 0 | 2
  Month 6: Much Worse | 12 | 3 | 2
  Month 6: Very Much Worse | 4 | 0 | 1
  Month 12: number analyzed (Participants) | 382 | 57 | 141
  Month 12: Very Much Improved | 93 | 9 | 32
  Month 12: Much Improved | 174 | 19 | 55
  Month 12: Minimally Improved | 80 | 20 | 28
  Month 12: Not Changed | 16 | 6 | 18
  Month 12: Minimally Worse | 7 | 1 | 2
  Month 12: Much Worse | 9 | 2 | 6
  Month 12: Very Much Worse | 3 | 0 | 0
  Month 18: number analyzed (Participants) | 304 | 73 | 139
  Month 18: Very Much Improved | 86 | 14 | 32
  Month 18: Much Improved | 136 | 34 | 55
  Month 18: Minimally Improved | 53 | 11 | 34
  Month 18: Not Changed | 14 | 10 | 11
  Month 18: Minimally Worse | 6 | 1 | 2
  Month 18: Much Worse | 7 | 2 | 5
  Month 18: Very Much Worse | 2 | 1 | 0
  Month 24: number analyzed (Participants) | 262 | 70 | 130
  Month 24: Very Much Improved | 93 | 10 | 34
  Month 24: Much Improved | 113 | 39 | 53
  Month 24: Minimally Improved | 34 | 10 | 27
  Month 24: Not Changed | 16 | 9 | 9
  Month 24: Minimally Worse | 5 | 2 | 2
  Month 24: Much Worse | 0 | 0 | 4
  Month 24: Very Much Worse | 1 | 0 | 1
  Month 30: number analyzed (Participants) | 214 | 64 | 143
  Month 30: Very Much Improved | 73 | 12 | 43
  Month 30: Much Improved | 102 | 41 | 63
  Month 30: Minimally Improved | 21 | 8 | 23
  Month 30: Not Changed | 12 | 2 | 12
  Month 30: Minimally Worse | 4 | 1 | 1
  Month 30: Much Worse | 1 | 0 | 1
  Month 30: Very Much Worse | 1 | 0 | 0
  Month 36: number analyzed (Participants) | 203 | 64 | 154
  Month 36: Very Much Improved | 85 | 22 | 53
  Month 36: Much Improved | 85 | 27 | 77
  Month 36: Minimally Improved | 22 | 9 | 15
  Month 36: Not Changed | 5 | 3 | 8
  Month 36: Minimally Worse | 1 | 1 | 1
  Month 36: Much Worse | 4 | 2 | 0
  Month 36: Very Much Worse | 1 | 0 | 0

60. Secondary Outcome: Number of Participants in Each Category of Clinical Global Impression-Tolerability (CGI-T) Scale at Month 3, 6, 12, 18, 24, 30 and 36
Description: CGI-T scale was a 7-point scale used to assess the tolerability of the study medication with respect to adverse events. Scale range/categories: 1= very high, 2= high, 3= above average, 4= average, 5= low, 6= very low, and 7= extremely low. Higher score indicated less tolerability with study medication.
Time Frame: Month 3, 6, 12, 18, 24, 30 and 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 546 | 65 | 96
Participants
  Month 3: number analyzed (Participants) | 546 | 2 | 96
  Month 3: Very High | 274 | 0 | 25
  Month 3: High | 123 | 0 | 18
  Month 3: Above Average | 40 | 0 | 18
  Month 3: Average | 69 | 2 | 30
  Month 3: Low | 22 | 0 | 3
  Month 3: Very Low | 10 | 0 | 2
  Month 3: Extremely Low | 8 | 0 | 0
  Month 6: number analyzed (Participants) | 468 | 29 | 95
  Month 6: Very High | 245 | 14 | 33
  Month 6: High | 116 | 4 | 12
  Month 6: Above Average | 28 | 1 | 20
  Month 6: Average | 49 | 6 | 23
  Month 6: Low | 19 | 2 | 2
  Month 6: Very Low | 5 | 1 | 4
  Month 6: Extremely Low | 6 | 1 | 1
  Month 12: number analyzed (Participants) | 367 | 52 | 74
  Month 12: Very High | 217 | 23 | 30
  Month 12: High | 84 | 12 | 14
  Month 12: Above Average | 19 | 3 | 12
  Month 12: Average | 35 | 10 | 14
  Month 12: Low | 11 | 4 | 4
  Month 12: Very Low | 1 | 0 | 0
  Month 12: Extremely Low | 0 | 0 | 0
  Month 18: number analyzed (Participants) | 298 | 64 | 69
  Month 18: Very High | 170 | 32 | 35
  Month 18: High | 77 | 15 | 9
  Month 18: Above Average | 16 | 3 | 7
  Month 18: Average | 26 | 10 | 11
  Month 18: Low | 5 | 3 | 6
  Month 18: Very Low | 2 | 0 | 0
  Month 18: Extremely Low | 2 | 1 | 1
  Month 24: number analyzed (Participants) | 250 | 65 | 60
  Month 24: Very High | 149 | 37 | 33
  Month 24: High | 67 | 17 | 12
  Month 24: Above Average | 9 | 5 | 3
  Month 24: Average | 19 | 3 | 8
  Month 24: Low | 4 | 3 | 4
  Month 24: Very Low | 2 | 0 | 0
  Month 24: Extremely Low | 0 | 0 | 0
  Month 30: number analyzed (Participants) | 210 | 59 | 57
  Month 30: Very High | 132 | 29 | 35
  Month 30: High | 55 | 18 | 5
  Month 30: Above Average | 7 | 6 | 6
  Month 30: Average | 12 | 5 | 9
  Month 30: Low | 2 | 1 | 1
  Month 30: Very Low | 1 | 0 | 1
  Month 30: Extremely Low | 1 | 0 | 0
  Month 36: number analyzed (Participants) | 197 | 56 | 58
  Month 36: Very High | 125 | 35 | 32
  Month 36: High | 51 | 12 | 10
  Month 36: Above Average | 11 | 3 | 6
  Month 36: Average | 7 | 5 | 7
  Month 36: Low | 0 | 1 | 2
  Month 36: Very Low | 1 | 0 | 0
  Month 36: Extremely Low | 2 | 0 | 1

61. Secondary Outcome: Number of Participants Who Were Responders According to Clinical Global Impression-Effectiveness (CGI-E) Scale at Month 3, 6, 12, 18, 24, 30 and 36
Description: The CGI-E was the value at which the participant's therapeutic benefit and adverse impact to the study drug intersected. Firstly clinician identified the degree of therapeutic benefit on scale range: very much improved, much improved, minimally improved, unchanged or worse. Secondly, the clinician rater identified the degree to which problems with tolerability adversely impact the participant on scale range: no adverse impact, mild adverse impact, moderate adverse impact, outweighs therapeutic effect. Finally, clinician identified in which participants benefits and adverse impacts intersected. Participants were then determined to be responders or non-responders to the study medication.
Time Frame: Month 3, 6, 12, 18, 24, 30 and 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 544 | 67 | 130
Participants
  Responders at Month 3: number analyzed (Participants) | 544 | 2 | 130
  Responders at Month 3 | 296 | 1 | 55
  Responders at Month 6: number analyzed (Participants) | 470 | 30 | 120
  Responders at Month 6 | 309 | 14 | 72
  Responders at Month 12: number analyzed (Participants) | 372 | 53 | 91
  Responders at Month 12 | 268 | 28 | 52
  Responders at Month 18: number analyzed (Participants) | 300 | 65 | 87
  Responders at Month 18 | 219 | 44 | 54
  Responders at Month 24: number analyzed (Participants) | 255 | 67 | 75
  Responders at Month 24 | 206 | 47 | 54
  Responders at Month 30: number analyzed (Participants) | 212 | 62 | 79
  Responders at Month 30 | 173 | 52 | 66
  Responders at Month 36: number analyzed (Participants) | 198 | 60 | 85
  Responders at Month 36 | 169 | 46 | 72

62. Secondary Outcome: Number of Participants in Each Category of Clinical Global Impression-Severity (CGI-S) Scale at Baseline, Month 3, 6, 12, 18, 24, 30 and 36
Description: CGI-S scale was a 7-point scale used to assess severity of illness on a range of 1 to 7; where, 1= normal, not mentally ill, 2= borderline mentally ill, 3= mildly mentally ill, 4= moderately mentally ill, 5= markedly mentally ill, 6= severely mentally ill, and 7= among the most extremely mentally. Higher score indicated worse condition.
Time Frame: Baseline, Month 3, 6, 12, 18, 24, 30 and 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 692 | 74 | 243
Participants
  Baseline: number analyzed (Participants) | 692 | 3 | 243
  Baseline: Normal, Not Mentally ill | 21 | 0 | 29
  Baseline: Borderline Mentally ill | 28 | 0 | 17
  Baseline: Mildly Mentally ill | 138 | 0 | 57
  Baseline: Moderately Mentally ill | 377 | 3 | 107
  Baseline: Markedly Mentally ill | 116 | 0 | 31
  Baseline: Severely Mentally ill | 12 | 0 | 2
  Baseline: Among the Most Extremely Mentally ill | 0 | 0 | 0
  Month 3: number analyzed (Participants) | 556 | 3 | 178
  Month 3: Normal, Not Mentally ill | 32 | 0 | 18
  Month 3: Borderline Mentally ill | 87 | 0 | 19
  Month 3: Mildly Mentally ill | 163 | 1 | 60
  Month 3: Moderately Mentally ill | 216 | 0 | 54
  Month 3: Markedly Mentally ill | 55 | 1 | 23
  Month 3: Severely Mentally ill | 3 | 1 | 4
  Month 3: Among the Most Extremely Mentally ill | 0 | 0 | 0
  Month 6: number analyzed (Participants) | 479 | 36 | 172
  Month 6: Normal, Not Mentally ill | 44 | 1 | 28
  Month 6: Borderline Mentally ill | 93 | 4 | 33
  Month 6: Mildly Mentally ill | 139 | 9 | 51
  Month 6: Moderately Mentally ill | 162 | 15 | 43
  Month 6: Markedly Mentally ill | 31 | 6 | 14
  Month 6: Severely Mentally ill | 10 | 1 | 3
  Month 6: Among the Most Extremely Mentally ill | 0 | 0 | 0
  Month 12: number analyzed (Participants) | 383 | 59 | 146
  Month 12: Normal, Not Mentally ill | 42 | 2 | 32
  Month 12: Borderline Mentally ill | 80 | 6 | 31
  Month 12: Mildly Mentally ill | 133 | 13 | 39
  Month 12: Moderately Mentally ill | 100 | 26 | 29
  Month 12: Markedly Mentally ill | 22 | 11 | 11
  Month 12: Severely Mentally ill | 6 | 1 | 4
  Month 12: Among the Most Extremely Mentally ill | 0 | 0 | 0
  Month 18: number analyzed (Participants) | 304 | 74 | 149
  Month 18: Normal, Not Mentally ill | 35 | 1 | 26
  Month 18: Borderline Mentally ill | 66 | 13 | 29
  Month 18: Mildly Mentally ill | 106 | 19 | 53
  Month 18: Moderately Mentally ill | 76 | 33 | 34
  Month 18: Markedly Mentally ill | 16 | 5 | 7
  Month 18: Severely Mentally ill | 5 | 3 | 0
  Month 18: Among the Most Extremely Mentally ill | 0 | 0 | 0
  Month 24: number analyzed (Participants) | 263 | 71 | 139
  Month 24: Normal, Not Mentally ill | 39 | 4 | 25
  Month 24: Borderline Mentally ill | 61 | 10 | 29
  Month 24: Mildly Mentally ill | 100 | 17 | 48
  Month 24: Moderately Mentally ill | 48 | 35 | 31
  Month 24: Markedly Mentally ill | 13 | 5 | 5
  Month 24: Severely Mentally ill | 2 | 0 | 1
  Month 24: Among the Most Extremely Mentally ill | 0 | 0 | 0
  Month 30: number analyzed (Participants) | 218 | 66 | 148
  Month 30: Normal, Not Mentally ill | 30 | 5 | 33
  Month 30: Borderline Mentally ill | 58 | 13 | 27
  Month 30: Mildly Mentally ill | 78 | 25 | 55
  Month 30: Moderately Mentally ill | 45 | 19 | 29
  Month 30: Markedly Mentally ill | 6 | 3 | 4
  Month 30: Severely Mentally ill | 1 | 1 | 0
  Month 30: Among the Most Extremely Mentally ill | 0 | 0 | 0
  Month 36: number analyzed (Participants) | 204 | 64 | 163
  Month 36: Normal, Not Mentally ill | 36 | 10 | 46
  Month 36: Borderline Mentally ill | 54 | 13 | 31
  Month 36: Mildly Mentally ill | 72 | 20 | 55
  Month 36: Moderately Mentally ill | 33 | 16 | 25
  Month 36: Markedly Mentally ill | 7 | 4 | 6
  Month 36: Severely Mentally ill | 2 | 1 | 0
  Month 36: Among the Most Extremely Mentally ill | 0 | 0 | 0

63. Secondary Outcome: Change From Baseline in Child Global Assessment Scale (CGAS) at Month 3, 6, 12, 18, 24, 30 and 36
Description: CGAS was to rate the general functioning of the study participants on a numeric scale of 1 to 100, where 1= extremely impaired and 100= doing very well.
Time Frame: Baseline, Month 3, 6, 12, 18, 24, 30 and 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 691 | 74 | 243
Units on scale
  Baseline: number analyzed (Participants) | 691 | 3 | 243
  Baseline | 55.80 (10.0) | 56.67 (5.8) | 59.86 (10.9)
  Change at Month 3: number analyzed (Participants) | 554 | 3 | 178
  Change at Month 3 | 6.58 (10.8) | -7.67 (8.7) | 4.61 (9.8)
  Change at Month 6: number analyzed (Participants) | 478 | 36 | 171
  Change at Month 6 | 8.24 (11.6) | 1.08 (16.5) | 8.23 (11.0)
  Change at Month 12: number analyzed (Participants) | 382 | 58 | 146
  Change at Month 12 | 10.02 (12.6) | 4.48 (9.4) | 10.66 (12.7)
  Change at Month 18: number analyzed (Participants) | 303 | 74 | 149
  Change at Month 18 | 10.51 (11.7) | 6.76 (10.5) | 12.46 (12.2)
  Change at Month 24: number analyzed (Participants) | 262 | 71 | 139
  Change at Month 24 | 11.29 (12.0) | 8.44 (11.3) | 11.29 (12.8)
  Change at Month 30: number analyzed (Participants) | 218 | 66 | 147
  Change at Month 30 | 12.37 (13.1) | 9.94 (11.4) | 12.54 (13.0)
  Change at Month 36: number analyzed (Participants) | 204 | 64 | 163
  Change at Month 36 | 13.05 (12.9) | 8.77 (10.7) | 15.28 (13.6)

64. Secondary Outcome: Change From Baseline in General Health and Social Functioning Using the Health of the Nation Outcome Scale for Children and Adolescents (HoNOSCA) Total Score at Month 3, 6, 12, 18, 24, 30 and 36
Description: HoNOSCA scale had 13-sub-scales used to assess general health and social functioning. 13 sub-scales were as the following: disruptive or aggressive behavior, attention deficit hyperactivity disorder (ADHD), self-harm, substance abuse, school problems, physical illness, psychosis, physical symptoms, internalizing symptoms, peer relationships, self-care, family relationships and school attendance problems. Each sub-scale had a range of 0 (no problems) to 4 (severe problems). Scores from all 13 sub-scales were summed up to give overall possible HoNOSCA total score range of 0 to 52. Higher score indicated worse condition.
Time Frame: Baseline, Month 3, 6, 12, 18, 24, 30 and 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Sertraline | Other Antidepressants | Psychotherapy
Number analyzed (Participants) | 685 | 72 | 241
Units on scale
  Baseline: number analyzed (Participants) | 685 | 3 | 241
  Baseline | 10.51 (5.4) | 8.33 (3.2) | 9.19 (4.6)
  Change at Month 3: number analyzed (Participants) | 542 | 3 | 172
  Change at Month 3 | -2.75 (4.8) | 4.33 (6.4) | -2.05 (4.2)
  Change at Month 6: number analyzed (Participants) | 469 | 36 | 169
  Change at Month 6 | -3.23 (5.1) | -0.14 (6.0) | -3.21 (4.7)
  Change at Month 12: number analyzed (Participants) | 377 | 59 | 144
  Change at Month 12 | -3.79 (5.5) | -2.46 (5.8) | -3.88 (4.8)
  Change at Month 18: number analyzed (Participants) | 298 | 72 | 144
  Change at Month 18 | -3.98 (5.6) | -3.53 (5.8) | -3.79 (4.6)
  Change at Month 24: number analyzed (Participants) | 257 | 69 | 136
  Change at Month 24 | -3.96 (5.4) | -5.07 (6.0) | -4.57 (4.7)
  Change at Month 30: number analyzed (Participants) | 210 | 65 | 147
  Change at Month 30 | -4.04 (4.8) | -4.75 (4.6) | -4.80 (5.1)
  Change at Month 36: number analyzed (Participants) | 201 | 62 | 162
  Change at Month 36 | -4.33 (5.3) | -4.69 (4.7) | -5.30 (5.1)

ADVERSE EVENTS:
Time Frame: Baseline up to 36 Months
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis population at each visit for respective arms was evaluated. Since participants switched from 1 treatment to another, hence at each visit participants analyzed were different from previous visit.
Groups:
- Sertraline (Baseline): Participants at Baseline (Day 1) or within 45 days of enrollment, initiated treatment with sertraline in routine clinical settings according to USPI provided by their physician.
- Other Antidepressants (Baseline): Use of other antidepressants at baseline was a study exclusion criterion, however, a few participants were enrolled who initiated treatment with an antidepressant.
- Psychotherapy (Baseline): Participants, 1) who were not taking sertraline or who failed a trial of sertraline judged adequate in dose and duration, and 2) initiated psychosocial rather than pharmacological treatment on or within 45 days of enrollment, for the same spectrum of mental health conditions that could have been treated with a SSRI medication.
- Sertraline (Month 3): Participants in this group were on sertraline only or sertraline and any other treatment at Month 3 visit.
- Other Antidepressants (Month 3): Participants in this group were on another antidepressant only or another antidepressant and psychotherapy at Month 3 visit.
- Psychotherapy (Month 3): Participants in this group were on psychotherapy only or no treatment at all at Month 3 visit.
- Sertraline (Month 6): Participants in this group were on sertraline only or sertraline and any other treatment at Month 6 visit.
- Other Antidepressants (Month 6): Participants in this group were on another antidepressant only or another antidepressant and psychotherapy at Month 6 visit.
- Psychotherapy (Month 6): Participants in this group were on psychotherapy only or no treatment at all at Month 6 visit.
- Sertraline (Month 12): Participants in this group were on sertraline only or sertraline and any other treatment at Month 12 visit.
- Other Antidepressants (Month 12): Participants in this group were on another antidepressant only or another antidepressant and psychotherapy at Month 12 visit.
- Psychotherapy (Month 12): Participants in this group were on psychotherapy only or no treatment at all at Month 12 visit.
- Sertraline (Month 18): Participants in this group were on sertraline only or sertraline and any other treatment at Month 18 visit.
- Other Antidepressants (Month 18): Participants in this group were on another antidepressant only or another antidepressant and psychotherapy at Month 18 visit.
- Psychotherapy (Month 18): Participants in this group were on psychotherapy only or no treatment at all at Month 18 visit.
- Sertraline (Month 24): Participants in this group were on sertraline only or sertraline and any other treatment at Month 24 visit.
- Other Antidepressants (Month 24): Participants in this group were on another antidepressant only or another antidepressant and psychotherapy at Month 24 visit.
- Psychotherapy (Month 24): Participants in this group were on psychotherapy only or no treatment at all at Month 24 visit.
- Sertraline (Month 30): Participants in this group were on sertraline only or sertraline and any other treatment at Month 30 visit.
- Other Antidepressants (Month 30): Participants in this group were on another antidepressant only or another antidepressant and psychotherapy at Month 30 visit.
- Psychotherapy (Month 30): Participants in this group were on psychotherapy only or no treatment at all at Month 30 visit.
- Sertraline (Month 36): Participants in this group were on sertraline only or sertraline and any other treatment at Month 36 visit.
- Other Antidepressants (Month 36): Participants in this group were on another antidepressant only or another antidepressant and psychotherapy at Month 36 visit.
- Psychotherapy (Month 36): Participants in this group were on psychotherapy only or no treatment at all at Month 36 visit.
Arm/Group | Sertraline (Baseline) | Other Antidepressants (Baseline) | Psychotherapy (Baseline) | Sertraline (Month 3) | Other Antidepressants (Month 3) | Psychotherapy (Month 3) | Sertraline (Month 6) | Other Antidepressants (Month 6) | Psychotherapy (Month 6) | Sertraline (Month 12) | Other Antidepressants (Month 12) | Psychotherapy (Month 12) | Sertraline (Month 18) | Other Antidepressants (Month 18) | Psychotherapy (Month 18) | Sertraline (Month 24) | Other Antidepressants (Month 24) | Psychotherapy (Month 24) | Sertraline (Month 30) | Other Antidepressants (Month 30) | Psychotherapy (Month 30) | Sertraline (Month 36) | Other Antidepressants (Month 36) | Psychotherapy (Month 36)
All-Cause Mortality (participants affected / at risk) | 0/614 | 0/3 | 0/181 | 0/622 | 0/19 | 0/384 | 0/516 | 0/48 | 0/181 | 0/426 | 0/80 | 0/181 | 0/335 | 0/84 | 0/181 | 0/289 | 0/83 | 0/181 | 1/240 | 0/85 | 0/181 | 0/207 | 0/73 | 0/181
Serious Adverse Events (participants affected / at risk) | 3/614 | 0/3 | 0/181 | 27/622 | 1/19 | 9/384 | 19/516 | 2/48 | 2/181 | 11/426 | 2/80 | 7/181 | 11/335 | 1/84 | 4/181 | 6/289 | 3/83 | 3/181 | 2/240 | 1/85 | 2/181 | 4/207 | 4/73 | 2/181
Other Adverse Events (participants affected / at risk) | 13/614 | 0/3 | 2/181 | 201/622 | 4/19 | 54/384 | 153/516 | 10/48 | 47/181 | 118/426 | 18/80 | 42/181 | 88/335 | 20/84 | 33/181 | 57/289 | 19/83 | 31/181 | 47/240 | 12/85 | 23/181 | 28/207 | 6/73 | 29/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sertraline (Baseline) (N=614) | Other Antidepressants (Baseline) (N=3) | Psychotherapy (Baseline) (N=181) | Sertraline (Month 3) (N=622) | Other Antidepressants (Month 3) (N=19) | Psychotherapy (Month 3) (N=384) | Sertraline (Month 6) (N=516) | Other Antidepressants (Month 6) (N=48) | Psychotherapy (Month 6) (N=181) | Sertraline (Month 12) (N=426) | Other Antidepressants (Month 12) (N=80) | Psychotherapy (Month 12) (N=181) | Sertraline (Month 18) (N=335) | Other Antidepressants (Month 18) (N=84) | Psychotherapy (Month 18) (N=181) | Sertraline (Month 24) (N=289) | Other Antidepressants (Month 24) (N=83) | Psychotherapy (Month 24) (N=181) | Sertraline (Month 30) (N=240) | Other Antidepressants (Month 30) (N=85) | Psychotherapy (Month 30) (N=181) | Sertraline (Month 36) (N=207) | Other Antidepressants (Month 36) (N=73) | Psychotherapy (Month 36) (N=181)
Drug ineffective (General disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anticholinergic syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Serotonin syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anger (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Emotional disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Homicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 0 | 7 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Self-injurious ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 4 | 1 | 3 | 4 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 10 | 1 | 6 | 9 | 1 | 2 | 5 | 0 | 4 | 6 | 1 | 3 | 4 | 3 | 3 | 1 | 1 | 2 | 3 | 3 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 4 | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Behaviour disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hostility (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sertraline (Baseline) (N=614) | Other Antidepressants (Baseline) (N=3) | Psychotherapy (Baseline) (N=181) | Sertraline (Month 3) (N=622) | Other Antidepressants (Month 3) (N=19) | Psychotherapy (Month 3) (N=384) | Sertraline (Month 6) (N=516) | Other Antidepressants (Month 6) (N=48) | Psychotherapy (Month 6) (N=181) | Sertraline (Month 12) (N=426) | Other Antidepressants (Month 12) (N=80) | Psychotherapy (Month 12) (N=181) | Sertraline (Month 18) (N=335) | Other Antidepressants (Month 18) (N=84) | Psychotherapy (Month 18) (N=181) | Sertraline (Month 24) (N=289) | Other Antidepressants (Month 24) (N=83) | Psychotherapy (Month 24) (N=181) | Sertraline (Month 30) (N=240) | Other Antidepressants (Month 30) (N=85) | Psychotherapy (Month 30) (N=181) | Sertraline (Month 36) (N=207) | Other Antidepressants (Month 36) (N=73) | Psychotherapy (Month 36) (N=181)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 9 | 0 | 3 | 11 | 1 | 5 | 5 | 1 | 3 | 3 | 1 | 2 | 4 | 1 | 2 | 3 | 0 | 1 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 6 | 0 | 4 | 9 | 0 | 2 | 3 | 0 | 2 | 3 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 4 | 1 | 5 | 6 | 0 | 0 | 4 | 0 | 2 | 6 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 6 | 0 | 3 | 3 | 0 | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 11 | 0 | 3 | 6 | 1 | 5 | 8 | 0 | 1 | 5 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 13 | 0 | 3 | 12 | 0 | 2 | 7 | 3 | 1 | 6 | 2 | 1 | 6 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 13 | 0 | 8 | 5 | 0 | 0 | 4 | 0 | 0 | 5 | 0 | 1 | 4 | 0 | 1 | 2 | 0 | 1 | 2 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 5 | 0 | 1 | 4 | 1 | 0 | 1 | 0 | 1 | 5 | 1 | 1 | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 26 | 1 | 8 | 33 | 0 | 8 | 19 | 1 | 9 | 15 | 4 | 5 | 14 | 4 | 8 | 4 | 1 | 1 | 8 | 0 | 4
Depressed mood (Psychiatric disorders) | 3 | 0 | 1 | 23 | 0 | 8 | 11 | 0 | 5 | 14 | 0 | 4 | 9 | 5 | 4 | 4 | 5 | 5 | 7 | 0 | 5 | 5 | 2 | 4
Hostility (Psychiatric disorders) | 4 | 0 | 1 | 22 | 1 | 9 | 19 | 0 | 6 | 17 | 3 | 3 | 11 | 0 | 5 | 6 | 2 | 3 | 0 | 1 | 3 | 0 | 1 | 5
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 10 | 0 | 3 | 9 | 1 | 0 | 7 | 1 | 1 | 8 | 1 | 0 | 3 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 2
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 29 | 2 | 7 | 21 | 0 | 8 | 9 | 2 | 8 | 7 | 1 | 9 | 6 | 4 | 5 | 4 | 3 | 1 | 2 | 0 | 5
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Albright's disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intentional product misuse (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 4 | 0 | 4 | 1 | 1 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 3 | 2 | 0 | 2 | 4 | 0 | 2 | 3 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 5 | 0 | 2 | 3 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 12 | 0 | 6 | 7 | 0 | 9 | 10 | 1 | 3 | 8 | 1 | 1 | 3 | 1 | 2 | 3 | 3 | 2 | 3 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 19 | 0 | 9 | 16 | 2 | 6 | 6 | 1 | 3 | 4 | 2 | 1 | 7 | 1 | 1 | 2 | 2 | 2 | 2 | 0 | 3
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 0 | 11 | 0 | 4 | 8 | 0 | 5 | 7 | 1 | 4 | 4 | 1 | 3 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 11 | 0 | 3 | 10 | 0 | 0 | 3 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 1
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blunted affect (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Compulsions (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dermatillomania (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enuresis (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Frustration tolerance decreased (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impulsive behaviour (Psychiatric disorders) | 0 | 0 | 0 | 4 | 0 | 2 | 10 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 1
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 0 | 10 | 0 | 0 | 15 | 0 | 1 | 9 | 0 | 2 | 6 | 2 | 0 | 4 | 1 | 0 | 4 | 0 | 2 | 2 | 2 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Social avoidant behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 10 | 0 | 2 | 8 | 2 | 3 | 7 | 1 | 2 | 1 | 2 | 4 | 3 | 0 | 1 | 2 | 0 | 3 | 2 | 0 | 1
Tachyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tic (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Trichotillomania (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Violence-related symptom (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 0 | 3 | 2 | 0 | 1 | 6 | 0 | 0 | 3 | 0 | 2 | 1 | 0 | 1 | 4 | 0 | 0 | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Obsessive-compulsive symptom (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oppositional defiant disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Self-injurious ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thinking abnormal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug ineffective (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Treatment noncompliance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Antisocial behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Communication disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Emotional distress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purging (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fight in school (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling jittery (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mononucleosis syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Defiant behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disinhibition (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Emotional disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Learning disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obsessive thoughts (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Precocious puberty (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sleep terror (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Attention-seeking behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Behaviour disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucinations, mixed (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT01302080/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT01302080/SAP_001.pdf